CLINICAL TRIAL: NCT00035256
Title: Sequential Use of Teriparatide and Raloxifene HCl in the Treatment of Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5490; B3D-MC-GHBQ
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2007-05-15 (Estimated); Status verified 2007-05

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Teriparatide; Raloxifene Hydrochloride

INTERVENTIONS:
Drug: teriparatide
Drug: raloxifene HCl
Drug: placebo

SUMMARY:
The purpose of this study is to determine whether the increase in spine bone mineral density that has been generally observed in previous clinical studies involving the study drug can be maintained or even increased if followed with raloxifene HCl. All qualifying study participants will receive the study drug followed by treatment with raloxifene HCl or placebo. All study participants will receive raloxifene HCl in the third phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with osteoporosis
* Must be female, age 55 through 80
* Must be at least 5 years postmenopausal
* Must be free of other severe or chronically disabling conditions
* Must be able to properly use injection device.

Exclusion Criteria:

* Must not have bone diseases other than osteoporosis
* Must not have history of certain cancers
* Must not have certain medical diseases (inflammatory bowel disease, malabsorption syndrome, kidney or bladder stones, venous thrombi or emboli, recent vaginal bleeding due to unknown causes)
* Must not have treatment with particular medications (warfarin, estrogens, androgens, steroids, calcitonins, fluorides, biphosphonates)
* Must not have known allergy to the study agent or raloxifene HCl

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Start 2001-10; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The study is designed to compare the effect of 1 year of raloxifene treatment with the effect of placebo on maintaining teriparatide-induced increases in spine and hip BMD.

SECONDARY OUTCOMES:
An open-label treatment phase will extend the study for 1 year beyond the primary endpoint. During this final year of the study all patients will receive raloxifene.
The purpose of lengthening is to assess the differences in response to raloxifene when it is administered immediately following versus 1 year after(with and without a washout period) withdrawal from teriparatide.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Maywood, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Portland, Oregon
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sainte-Foy, Quebec